CLINICAL TRIAL: NCT05205772
Title: Investigating Central Neurophysiologic Correlates of Non-Motor Symptoms of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-0751
Record Dates: First submitted 2021-12-02; First posted 2022-01-25 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Autonomic Dysfunction; Depression
MeSH Terms: conditions — Parkinson Disease; Primary Dysautonomias; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded as to which site is being stimulated, experimental site or control site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- medial prefrontal cortex - control site - dorsolateral prefrontal cortex (Experimental): Participants first undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex.
  Interventions: Device: transcranial magnetic stimulation
- medial prefrontal cortex - dorsolateral prefrontal cortex - control site (Experimental): Participants first undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the control site.
  Interventions: Device: transcranial magnetic stimulation
- dorsolateral prefrontal cortex - medial prefrontal cortex - control site (Experimental): Participants first undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the control site.
  Interventions: Device: transcranial magnetic stimulation
- dorsolateral prefrontal cortex - control site - medial prefrontal cortex (Experimental): Participants first undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the medial prefrontal cortex.
  Interventions: Device: transcranial magnetic stimulation
- control site - medial prefrontal cortex - dorsolateral prefrontal cortex (Experimental): Participants first undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex.
  Interventions: Device: transcranial magnetic stimulation
- control site - dorsolateral prefrontal cortex - medial prefrontal cortex (Experimental): Participants first undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the medial prefrontal cortex.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
  Other Names: intermittent theta-burst stimulation (iTBS)

SUMMARY:
This is a randomized, single-blinded, triple crossover study focused on determining the feasibility of using transcranial magnetic stimulation (TMS) for treatment of Parkinson's disease related autonomic dysfunction and depression. Participants will undergo TMS to three brain regions: medial prefrontal cortex (mPFC) (experimental site), dorsolateral prefrontal cortex (DLPFC) (alternative experimental site), or primary sensory cortex (S1) (control site) in a triple crossover design. Participants will complete symptom questionnaires, neurologic examination and cognitive assessments, and orthostatic vital signs recording before and after each brain stimulation session.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 50 and 90 years of age, without a diagnosis of severe dementia
* Carry a diagnosis of idiopathic Parkinson's disease based on the United Kingdom Parkinson's Disease Society Brain Bank clinical diagnostic criteria
* Have had symptoms of Parkinson's disease for at least 3 years
* Hospital's study-specific informed consent must be obtained
* Must have capacity to provide informed consent in English
* For female participants, confirmation that a menstrual period has not occurred in over 12 months, or that an effective form of contraception will be used during the study

Exclusion Criteria:

* Inability to provide informed consent.
* Severe dementia
* History of epilepsy or brain surgery
* Severe tremor or dyskinesia that would interfere with EEG as determined by the PI
* Parkinson's patients with clinically significant medical or neurological conditions which may be an alternative cause of orthostatic hypotension, such as neuropathy, renal failure, heart failure, cardiac arrhythmias, severe diabetes, or spinal cord injuries
* The investigators will exclude patients who are treated with medications which can significantly lower blood pressure or heart rate, such as antihypertensive medications, diuretics, and alpha-blocking medications
* Presence of other known central nervous system disease that may interfere with performance or interpretation of EEG or TMS
* Presence of any implanted metal devices including, but not limited to, pacemakers, deep brain stimulators, vagal nerve stimulators, bladder stimulators, or cochlear implants.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Sklerov, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 months to 36 months after publication.
Access Criteria: Data will be made available to investigators who have approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex: Participants first undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex.
  transcranial magnetic stimulation: Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  Intermittent theta-burst stimulation (iTBS) is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site: Participants first undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the control site.
  transcranial magnetic stimulation: Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site: Participants first undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the control site.
  transcranial magnetic stimulation: Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex: Participants first undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the medial prefrontal cortex.
  transcranial magnetic stimulation: Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex: Participants first undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex.
  transcranial magnetic stimulation: Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex: Participants first undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the medial prefrontal cortex.
  transcranial magnetic stimulation: Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
Period: Screening
Arm/Group | Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex | Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex | Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex | Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex
Started | 5 | 4 | 5 | 3 | 7 | 6
Completed | 5 | 4 | 5 | 3 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention
Arm/Group | Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex | Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex | Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex | Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex
Started | 5 | 3 | 5 | 3 | 7 | 5
Completed | 5 | 2 | 5 | 2 | 6 | 5
Not Completed | 0 | 1 | 0 | 1 | 1 | 0
Period: Washout (3 Weeks)
Arm/Group | Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex | Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex | Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex | Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex
Started | 5 | 2 | 5 | 2 | 6 | 5
Completed | 5 | 2 | 4 | 2 | 6 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex | Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex | Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex | Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex
Started | 5 | 2 | 4 | 2 | 6 | 5
Completed | 5 | 2 | 4 | 2 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (3 Weeks)
Arm/Group | Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex | Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex | Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex | Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex
Started | 5 | 2 | 4 | 2 | 6 | 5
Completed | 5 | 2 | 4 | 2 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex | Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex | Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex | Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex
Started | 5 | 2 | 4 | 2 | 6 | 5
Completed | 5 | 2 | 4 | 2 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex: Participants first undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the control site. After a 3 week washout period, participants undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex.
  transcranial magnetic stimulation: Transcranial magnetic stimulation (or TMS) is a non-invasive form of brain stimulation in which a magnetic pulse is applied directly to the scalp. This device is FDA approved for treatment of depression and other neuropsychiatric disorders, and is regularly used in neurologic and psychiatric research.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Total: Total of all reporting groups
Arm/Group | Medial Prefrontal Cortex - Control Site - Dorsolateral Prefrontal Cortex | Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex - Control Site | Dorsolateral Prefrontal Cortex - Control Site - Medial Prefrontal Cortex | Control Site - Medial Prefrontal Cortex - Dorsolateral Prefrontal Cortex | Control Site - Dorsolateral Prefrontal Cortex - Medial Prefrontal Cortex | Total
Number analyzed (Participants) | 5 | 2 | 4 | 2 | 6 | 5 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.36) | 68.5 (7.50) | 69.5 (3.77) | 74.0 (1.00) | 67.0 (9.27) | 67.2 (8.73) | 67.92 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 1 | 2 | 10
  Male | 3 | 0 | 3 | 0 | 5 | 3 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 4 | 2 | 6 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Frontal Midline Theta EEG Power After Brain Stimulation
Description: Degree of change of frontal midline theta (FMT) power on electroencephalography (EEG) after brain stimulation at each site (medial prefrontal cortex, dorsolateral prefrontal cortex, control site).
Time Frame: At least 30 minutes before initial iTBS, and 30 minutes after each iTBS treatment
Population: Data are reported for participants who completed all 3 treatment interventions.
Measure: Mean (Standard Deviation); unit: microvolts^2/Hz
Groups:
- Medial Prefrontal Cortex Stimulation: Participants received transcranial magnetic stimulation to the medial prefrontal cortex.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Dorsolateral Prefrontal Cortex Stimulation: Participants received transcranial magnetic stimulation to the dorsolateral prefrontal cortex.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
- Control Site Stimulation: Participants first undergo transcranial magnetic stimulation to the dorsolateral prefrontal cortex. After a 3 week washout period, participants then undergo transcranial magnetic stimulation to the medial prefrontal cortex. After a 3 week washout period, Participants received transcranial magnetic stimulation to the control site.
  iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes.
Arm/Group | Medial Prefrontal Cortex Stimulation | Dorsolateral Prefrontal Cortex Stimulation | Control Site Stimulation
Number analyzed (Participants) | 24 | 24 | 24
microvolts^2/Hz | 1.03 (2.41) | 0.44 (2.55) | 1.01 (2.13)
Statistical Analysis 1: Comparison: Medial Prefrontal Cortex Stimulation; Test type: Other; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dorsolateral Prefrontal Cortex Stimulation; Test type: Other; p = 0.54, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Site Stimulation; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Medial Prefrontal Cortex Stimulation vs Control Site Stimulation; Test type: Superiority; p = 0.98, ANOVA
Statistical Analysis 5: Comparison: Dorsolateral Prefrontal Cortex Stimulation vs Control Site Stimulation; Test type: Superiority; p = 0.41, ANOVA
Statistical Analysis 6: Comparison: Medial Prefrontal Cortex Stimulation vs Dorsolateral Prefrontal Cortex Stimulation vs Control Site Stimulation; Test type: Superiority; p = 0.63, ANOVA

2. Primary Outcome: Correlation Between the Scales for Outcomes in Parkinson's Disease - Autonomic (SCOPA-AUT) Total Score and EEG
Description: Degree of correlation between the Scales for Outcomes in Parkinson's disease - Autonomic (SCOPA-AUT) total score and frontal midline theta EEG power extracted from Baseline pre-stimulation initial visit EEG and SCOPA-AUT questionnaire. The SCOPA-AUT is a validated autonomic symptom survey for people with Parkinson's disease. It contains 6 domains (gastrointestinal, urinary, cardiovascular, thermoregulatory, pupillary, and sexual). The investigators will use the total composite score including all domains. The score range is 0-69, with a total of 23 questions. 0 means no symptoms, 69 is highest burden of symptoms. The FMT and SCOPA-AUT were assessed at baseline. FMT power and SCOPA-AUT were correlated using the Spearman Correlation Coefficient calculation. A positive correlation coefficient indicates a positive relationship between the assessments; higher FMT power correlates with higher symptom burden.
Time Frame: At least 30 minutes before initial iTBS
Measure: Number; unit: Spearman Correlation coefficient
Groups:
- Stimulation Naiive: All participants prior to first stimulation.
Arm/Group | Stimulation Naiive
Number analyzed (Participants) | 24
Spearman Correlation coefficient | 0.255
Statistical Analysis 1: Comparison: Stimulation Naiive; Test type: Other; p = 0.38, Regression, Linear — Adjusted for age

3. Primary Outcome: Correlation Between the Orthostatic Hypotension Questionnaire (OHQ) and EEG
Description: Degree of correlation between the Orthostatic Hypotension Questionnaire (OHQ) composite score and frontal midline theta EEG power extracted from Baseline pre-stimulation initial visit EEG and OHQ questionnaire. The OHQ consists of two sections: 1-orthostatic hypotension symptom assessment, which includes 6 questions with a score range of 0-66 (0 is no symptoms, 66 is most severe symptoms); and 2-the orthostatic hypotension daily activity scale, which rates interference of symptoms on activities of daily living. This part consists of four questions, and score range is 0-44 (0 is no interference, 44 is most severe interference). The composite OHQ score is the average score between these two subsections. FMT power and OHQ were correlated using the Spearman Correlation Coefficient calculation. A positive correlation coefficient indicates a positive relationship between the assessments; higher FMT power correlates with higher symptom burden.
Time Frame: At least 30 minutes before initial iTBS
Measure: Number; unit: Spearman Correlation coefficient
Arm/Group | Stimulation Naiive
Number analyzed (Participants) | 24
Spearman Correlation coefficient | 0.261
Statistical Analysis 1: Comparison: Stimulation Naiive; Test type: Other; p = 0.67, Regression, Linear — Adjusted for age

4. Primary Outcome: Correlation Between Degree of Orthostatic Hypotension and EEG
Description: Degree of correlation between degree of orthostatic hypotension and frontal midline theta EEG power will be measured extracted from Baseline pre-stimulation visit EEG and blood pressure measures. Orthostatic vital signs will be measured at least 30 minutes before initial iTBS as follows: blood pressure will be measured after at least 3 minutes of rest in the supine position. Blood pressure will again be measured after 3 minutes of standing. Blood pressure reduction is expressed as the magnitude of reduction, thus a positive number reflects a greater reduction. Lack of blood pressure reduction was coded as '0'. A positive correlation coefficient indicates a positive relationship between the assessments; higher FMT power correlates with higher more severe orthostatic hypotension.
Time Frame: At least 30 minutes before initial iTBS
Measure: Number; unit: Spearman Correlation coefficient
Arm/Group | Stimulation Naiive
Number analyzed (Participants) | 24
Spearman Correlation coefficient | 0.429
Statistical Analysis 1: Comparison: Stimulation Naiive; Test type: Other; p = 0.156, Regression, Linear

5. Other Pre Specified Outcome: SCOPA-AUT Response to Brain Stimulation
Description: Change in the SCales for Outcomes in Parkinson's disease - Autonomic (SCOPA-AUT) from 30 minutes before stimulation to 1 day after stimulation and 4 days after stimulation. The SCOPA-AUT is a validated autonomic symptom survey for people with Parkinson's disease. It contains 6 domains (gastrointestinal, urinary, cardiovascular, thermoregulatory, pupillary, and sexual). The investigators will use the total composite score including all domains. The score range is 0-69, with a total of 23 questions. 0 means no symptoms, 69 is highest burden of symptoms
Time Frame: 30 minutes pre-iTBS, and 1 day and 4 days after each iTBS treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: OHQ Response to Brain Stimulation
Description: Change in the Orthostatic Hypotension Questionnaire (OHQ) from before to after iTBS. The OHQ will be administered at least 30 minutes before stimulation, and again 1 day and 4 days after stimulation. The OHQ is an orthostatic hypotension symptom survey and consists of two sections. The first is the orthostatic hypotension symptom assessment, which includes 6 questions with a score range of 0-66 (0 is no symptoms, 66 is most severe symptoms). The second part is the orthostatic hypotension daily activity scale, which rates interference of symptoms on activities of daily living. This part consists of four questions, and score range is 0-44 (0 is no interference, 44 is most severe interference). The investigators will calculate the composite OHQ score, which is the average score between these two subsections.
Time Frame: At least 30 minutes pre-iTBS, and day 1 and day 4 after each iTBS treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Response of Orthostatic Blood Pressure Changes to Brain Stimulation
Description: Change in the orthostatic blood pressure change from before to after iTBS. Orthostatic vital signs will be measured as follows: blood pressure will be measured after at least 3 minutes of rest in the supine position. Blood pressure will again be measured after 3 minutes of standing. This will be measured at least 30 minutes before brain stimulation, and again 30 minutes after brain stimulation.
Time Frame: At least 30 minutes before each iTBS treatment, and 30 minutes after each iTBS treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Depression Symptom Response to Brain Stimulation
Description: Change in the Beck Depression Inventory II (BDI-II) from before to after iTBS. Participants will complete the BDI-II at least 30 minutes before brain stimulation. The questionnaire will be repeated 1 day and 4 days after stimulation. The BDI-II is a validated depression symptom survey. This survey contains 21 questions, with a score range of 0-63, where 0 means no depression symptoms and 63 indicates severe depression symptoms.
Time Frame: At least 30 minutes before each iTBS treatment, and day 1 and day 4 after each iTBS treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 1-3 days following completion of the 3rd intervention, approximately 6-7 weeks total depending upon optional consolidation of screening and Visit 1 as per protocol.
Arm/Group | Medial Prefrontal Cortex Stimulation | Dorsolateral Prefrontal Cortex Stimulation | Control Site Stimulation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 1/26 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medial Prefrontal Cortex Stimulation (N=25) | Dorsolateral Prefrontal Cortex Stimulation (N=26) | Control Site Stimulation (N=25)
Hair Loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exacerbation of Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT05205772/Prot_SAP_000.pdf